CLINICAL TRIAL: NCT07221968
Title: Melatonin for the Treatment of Developmental/Epileptic Encephalopathy With Spike Wave Activation In Sleep (DEE-SWAS; Formerly ESES)
Brief Title: Melatonin for the Treatment of DEE-SWAS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Carosella, Christopher, Assistant Professor of Neurology, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00478764
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: CSWS; Developmental and/or Epileptic Encephalopathies; Electrical Status Epilepticus in Sleep
Keywords: DEE-SWAS; ESES; CSWS; epileptic encephalopathy; melatonin
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Single dose administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Melatonin (Experimental): Melatonin 0.3mg/kg (20mg max)
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Melatonin will be used in single fixed dose as described

SUMMARY:
The goal of this study is to learn if melatonin, a naturally produced substance, can help to treat some of the symptoms of DEE-SWAS, a type of epilepsy that causes children to lose skills and development. It will look at doses of melatonin that are higher than most people use.

The study will look at the safety of melatonin in patients with DEE-SWAS The study will look at the ways melatonin affects abnormal brain activity on a study called an EEG.

The study will look at the ways melatonin affects normal brain activity that occurs in sleep.

ELIGIBILITY:
Inclusion Criteria:

Clinic Dx of DEE-SWAS

1. Dx of DEE-SWAS by a board-certified pediatric neurology/epileptologist Clinical history of delayed milestones in at least 1 category, regression of milestones in at least 1 category, and/or failure to progress in milestones in at least 1 category
2. Abnormal baseline neuropsychiatric testing consistent with Dx Abnormal EEG
3. Epileptiform abnormalities (spike, polyspike, sharp) in at least 1 head region
4. Increase by 2-fold of epileptiform abnormalities during NREM sleep as compared to wakefulness
5. SWI of ≥50% in at least one head region on overnight EEG

Exclusion Criteria:

1. Allergic to ingredients in study drug Melatonin

   * Hypoallergenic plant fiber (cellulose)
   * Active use of the medication viloxazine
2. History of known cardiac rhythm abnormalities, heart failure or decreased EF <30%
3. History of known pulm requiring oxygen or invasive positive pressure ventilation. Patients with non-invasive PPV (e.g. CPAP) due OSA w/o 02 requirement, rate, or DX of CSA, on stable pressure settings for >3 mnths will not be excluded.
4. History of liver dysf OR AST/ALT/AlkPhos >2.5 ULN w/i year. If lab value meeting exclusion between 3-12 months, a repeat lab value < 2.5 ULN will be considered for inclusion
5. Post-menarchal participants. of childbearing potential with a positive urine pregnancy test

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Within 24 hours of dose administration
  This study will evaluate for adverse events associated with single high dose melatonin administration
Side effects | Within 24 hours of dose administration
  This study will evaluate for multiorgan adverse effects associated with single high dose melatonin administration based on standardized questionnaire assessment. The assessment is a multiorgan adverse event questionnaire described in Jarernsiripornkul 2001, modified to reflect single dosing rather than chronic dosing. The results of this questionanaire are descriptive.

SECONDARY OUTCOMES:
Spike wave index (SWI) | Within 24 hours of dose administration
  This study will evaluate change in epileptiform activity during NREM sleep as defined by common clinical definition of SWI - average percentage of second bins containing an epileptiform discharge during NREM sleep
Sleep spindle | Within 24 hours of dose administration
  This study will evaluate change in sleep spindle activity during NREM sleep using both blinded review and validated deep learning algorithmic detection.
Salivary melatonin pharmacokinetics | 24 hours prior to intervention and 24 hours following intervention
  Baseline and post intervention salivary melatonin levels will be obtained at multiple time points

IPD SHARING:
Plan to Share IPD: Undecided